CLINICAL TRIAL: NCT05808660
Title: Questionable Health Behaviors and Their Distal and Proximal Correlates: Protocol for a Nationally Representative Survey in Serbia
Brief Title: Questionable Health Behaviors and Their Distal and Proximal Correlates
Acronym: REASON4HEALTH
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Ljiljana Lazarevic, Senior Researcher, University of Belgrade
Other Study IDs: 7739597; 7739597 (Other Grant/Funding Number: Science Fund of the Republic of Serbia)
Record Dates: First submitted 2023-03-28; First posted 2023-04-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Questionable Health Behaviors and Their Distal and Proximal Correlates
Keywords: TCAM/ iNAR/ distal predictors /proximal predictors / irrational mindset

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population

SUMMARY:
The goals of the study:

1. to investigate the frequency of Traditional, Complementary and Alternative Medicine use (TCAM) and intentional Non-adherence to medical recommendations (iNAR) in the general population in Serbia, as well as their mutual relations.
2. to examine the distribution of irrational beliefs in the general population;
3. to explore the relationships between TCAM and iNAR behaviors on the one hand and variables of personality, thinking styles and cognitive reflection on the other, with a major assumption that these relationships will be mediated by the domain of irrational beliefs and socio-political attitudes.

Participants will respond to a battery of instruments assessing TCAM use and iNAR, as well as, sociodemographics and health-related variables (such as health status, chronic diseases, BMI, etc.), distal psychological (i.e. personality, thinking disposition and styles) and proximal psychological, variables, (i.e. the irrational mindset, as well as socio-political beliefs and attitudes).

Data will be collected on the probabilistic household sample representative for the general population in Serbia (N=1043).

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years of age

Exclusion Criteria:

* the inability to understand the Serbian language
* failure to pass any of the four attention-check questions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Traditional, complementary and alternative medicine (TCAM) use | baseline
  Prevalence of TCAM use
intentional non-adherence to official medical recommendations (iNAR) | baseline
  Prevalence of iNAR

CONTACTS AND LOCATIONS:
Overall Officials: Goran Knezevic, prof., Principal Investigator — Department of Psychology, Faculty of Philosophy, University of Belgrade
Locations (1):
- Faculty of Philosophy, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knezevic G, Lazarevic L, Puric D, Zupan Z, Zezelj I. Prevalence of questionable health behaviours in Serbia and their psychological roots: protocol for a nationally representative survey. BMJ Open. 2023 Oct 12;13(10):e075274. doi: 10.1136/bmjopen-2023-075274. PMID 37827738